CLINICAL TRIAL: NCT01209403
Title: Insulin-like Growth Factor (IGF-I) in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IGFHD1-2010; 2010-020114-29 (EudraCT Number)
Record Dates: First submitted 2010-09-17; First posted 2010-09-27 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Kidney Failure, Chronic
Keywords: Dialysis; Malnutrition; Insulin-Like Growth Factor I; Insulin-Like Growth Factor Binding Protein 1; Inflammation
MeSH Terms: conditions — Kidney Failure, Chronic; Malnutrition; Inflammation | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No treatment (No Intervention)
- Glukose-infusion (Active Comparator): Glucose-infusion during hemodialysis
  Interventions: Drug: Glucose-infusion
- Glucose-insulin infusion (Active Comparator): Glucose-insulin infusion during hemodialysis
  Interventions: Drug: Glucose-insulin infusion

INTERVENTIONS:
Drug: Glucose-infusion — Continuous iv infusion of glucose
  Other Names: Glukose
  Arms: Glukose-infusion
Drug: Glucose-insulin infusion — Continuous iv infusion of glucose and shortlasting
  Other Names: Glukose; Novorapid
  Arms: Glucose-insulin infusion

SUMMARY:
The purpose of this study is to investigate whether the anabolic potentials of insulin may be used to reverse the catabolic effects of hemodialysis in non-diabetic patients with end-stage renal failure.

DETAILED DESCRIPTION:
Nutritional markers such as lean body mass and serum albumin are strong predictors of the mortality and morbidity in patients with end-stage renal failure (ESRF) on maintenance hemodialysis (HD). Maintenance HD is considered to contribute to the malnutrition of patients with ESRF, but the exact mechanism has remained unknown. However, we have recently shown that the bioactivity of insulin-like growth factor-I (IGF-I) is reduced by 50% during HD. Furthermore, we showed that the reduction in the bioactivity of IGF-I is directly linked to an up-regulation of IGF-binding protein-1 (IGFBP-1), the only acutely regulated IGFBP, which increased by 6-fold during HD. IGFBP-1 is produced in the liver, primarily under the control of insulin, which promptly inhibits the hepatic production of IGFBP-1. As plasma insulin remains fairly low during a maintenance HD, the increase in IGFBP-1 may be explained by the absence of insulin.

The finding that HD acutely down-regulates the bioactivity of IGF-I by an up-regulation of IGFBP-1 may not only explain the catabolic mechanisms of HD per se, it also opens for a new treatment strategy of ESRF patients undergoing maintenance HD. Thus, on the basis of our previous study we hypothesize that treatment of ERSF patients with high doses of insulin during maintenance HD may counter-act the HD-induced stimulation of IGFBP-1, making it possible to preserve the bioactivity of IGF-I, and thereby abolishing the catabolic impact of HD.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* stable patients on maintenance hemodialysis for > 3 months
* well-functioning arteriovenous (AV) shunt with recirculation < 5%
* informed consent

Exclusion Criteria:

* diabetes mellitus
* body mass index < 18.5 kg/m2 or > 30 kg/m2
* malnutrition (subjective global assessment (SGA) score C)
* malignancy
* use of immunosuppressive drugs including glucocorticosteroids
* severe infectious disease < 4 weeks
* pregnancy

Exclusion Criteria during the study:

* myocardial infarction or arrythmia with hemodynamic derangements
* permanent thrombosis in the arteriovenous (AV) shunt
* severe infectious disease
* renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Effect of glucose and glucose-insulin infusion on plasma IGF-I and IGFBP-1 during hemodialysis | From 2 h prior to start of hemodialysis to 2 h after end of hemodialysis
  All patients are randomly assigned to a hemodialysis session with either i) no infusion, ii) a continuous iv infusion of glucose, and iii) a continuous iv infusion of glucose and shortacting insulin. Each dialysis session will be separated by 2 weeks of wash-out

SECONDARY OUTCOMES:
Relationship between inflammatory markers and plasma concentrations of IGF-I and IGFBP-1 during hemodialysis | From 2 h prior to start of hemodialysis to 2 h after end of hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Per Ivarsen, MD, PhD, Study Director — Department of Nephrology, Aarhus University Hospital, Skejby; Jan Frystyk, MD,PhD,DMSc, Study Director — Department of Endocrinology and Internal Medicine, Aarhus University Hospital; Bente Jespersen, MD, DMSc, Study Director — Department of Nephrology, Aarhus University Hospital, Skejby; Mark Reinhard, MD, Principal Investigator — Department of Nephrology, Aarhus University Hospital, Skejby
Locations (1):
- Department of Nephrology, Aarhus University Hospital, Skejby, Aarhus, Denmark

REFERENCES:
- [Derived] Reinhard M, Frystyk J, Jespersen B, Bjerre M, Christiansen JS, Flyvbjerg A, Ivarsen P. Effect of hyperinsulinemia during hemodialysis on the insulin-like growth factor system and inflammatory biomarkers: a randomized open-label crossover study. BMC Nephrol. 2013 Apr 4;14:80. doi: 10.1186/1471-2369-14-80. PMID 23557110